CLINICAL TRIAL: NCT05730400
Title: Histological Assessment of Deproteinized Bovine Bone Loaded by Bone Marrow Aspirate Versus Deproteinized Bovine Bone Alone for Guided Sinus Floor Elevation. (A Randomized Controlled Clinical Trial)
Brief Title: Histological Assessment of BMAC Utilized in Sinus Lift
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Walaa Kadry, Lecturer of oral and Maxillofacial Surgery, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BMAC for sinus augmentation
Record Dates: First submitted 2023-01-26; First posted 2023-02-15 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Implant Site Reaction
Keywords: Bone marrow; Sinus augmentation; Sinus lift

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BMAC/bovine graft (Active Comparator): Bone marrow aspirate concentrate loaded on bovine graft (Tutogen Medical GmbH, Neunkirchen am Brand, Germany, 1- 2mm particle size) utilization for sinus floor augmentation with residual alveolar bone height less than 5 mm, 1st arm
  Interventions: Drug: BMAC loaded on bovine graft
- Bovine graft group (Active Comparator): bovine graft utilization for sinus floor augmentation with residual alveolar bone height less than 5 mm, 2nd arm
  Interventions: Drug: Bovine graft only

INTERVENTIONS:
Drug: BMAC loaded on bovine graft — Bone marrow aspirate concentrate loaded on bovine graft for sinus floor augmentation
  Other Names: Bone marrow aspirate concentrate loaded on bovine graft
  Arms: BMAC/bovine graft
Drug: Bovine graft only — Bovine graft only for sinus floor augmentation
  Other Names: Unloaded bovine graft
  Arms: Bovine graft group

SUMMARY:
Aim : The aim of present study was to evaluate BMAC/bovine graft utilization in Sinus membrane augmentation on bone quality and quantity. Methodology: sixteen patients suffering from atrophic posterior maxilla with sinus pneumatization were randomly divided into two equal groups: study group: the sinus membrane was elevated with BMAC/bovine graft whereas the control group recieved bovine graft only for sinus floor augmentation.

All patients will be evaluated at 1 week, 4 months to measure bone height and bone core biopsy for histological assessment at 4 months during implant placement.

DETAILED DESCRIPTION:
Aim : The aim of present study was to evaluate BMAC/bovine graft utilization in Sinus membrane augmentation on bone height gain and quality of bone on histological assessment.

Methodology: sixteen patients suffering from atrophic posterior maxilla with sinus pneumatization were randomly divided into two equal groups: study group: the sinus membrane was elevated with bone marrow aspirate concentrate loaded on bovine graft whereas the control group recieved bovine graft only for sinus floor augmentation.

All patients will be evaluated at 1 week, 4 months by CBCT to measure bone height and bone core biopsy for histological assessment at 4 months during implant placement.

ELIGIBILITY:
Inclusion Criteria:

* Patients with missing upper posterior teeth and atrophic posterior maxilla with a residual bone height ranging from 4 to 6 mm
* Patients who has as deficient as 4 mm vertical bone height in posterior maxilla that need bone augmentation before delayed implant placement.
* Highly motivated patients

Exclusion Criteria:

* Patients suffering from any systemic disease or those under any medication that may interfere with normal bone healing.
* Patients suffering from any sinus pathosis.
* Patients with conditions that could potentially compromise BM quality, previous BMA, or acute illness.
* Heavy smoker (> 20 cigarettes daily)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-10-30 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Histological assessment | After 4 months of surgery
  Histological assessment of core biopsy obtained at time of implant placement for percentage of new bone formation and residual graft

SECONDARY OUTCOMES:
Implant stability | After 4 months of surgery
  implant stability immediately following installation after 4 months using ostell device (ISQ scale)
Bone gain | Preoperative, immediate and 4 months Postoperative
  Vertical bone height gain from sinus floor on cone beam ct

CONTACTS AND LOCATIONS:
Overall Officials: Maha Hakam, Phd, Study Director — Professor at Faculty of Dentistry Cairo University
Locations (1):
- Faculty of Dentistry, department of oral and Maxillofacial Surgery, Cairo, Egypt